CLINICAL TRIAL: NCT04936880
Title: Pilot Study on the Evaluation of the Effectiveness of a Virtual Reality Device on Anxiety During Procedural Sedation in Traumatology in Emergency Department
Acronym: VIRTUAL DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIRTUAL DREAM
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-01

CONDITIONS: Reality Device; Reduction Procedure; Fracture; Dislocation
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : Virtual reality + analgesia-sedation (Experimental): Use of a virtual reality device + analgesia-sedation drugs according to SFMU/SFAR 2010 guidelines during reduction procedure
  Interventions: Device: Experimental : Virtual reality + analgesia-sedation
- Control: Analgesia-sedation (Active Comparator): Use of analgesia-sedation drugs according to SFMU/SFAR 2010 guidelines during reduction procedure
  Interventions: Drug: Control: Analgesia-sedation

INTERVENTIONS:
Device: Experimental : Virtual reality + analgesia-sedation — Use of a virtual reality device + analgesia-sedation drugs according to SFMU/SFAR 2010 guidelines during reduction procedure
  Arms: Experimental : Virtual reality + analgesia-sedation
Drug: Control: Analgesia-sedation — Use of analgesia-sedation drugs according to SFMU/SFAR 2010 guidelines during reduction procedure
  Arms: Control: Analgesia-sedation

SUMMARY:
The aim of this study is to evaluate the efficiency of a reality device and a virtual hypnosis software to reduce the anxiety during reduction procedure in traumatology in an emergency department. These devices have recently been evaluated in the management of pain and anxiety in different specialties but never in the context of analgesia-sedation protocols in emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient suffering from one of the following traumatic pathologies requiring a technical procedure in the emergency room Shoulder dislocation Ankle dislocation Elbow dislocation Wrist dislocation Reducible fractures
* No contraindication to Virtual Reality
* No contraindication to morphine, ketamine, propofol, paracetamol, nefopam and MEOPA
* Patient having given oral, free and informed consent

Exclusion Criteria:

* Patients suffering from mono or binocular blindness
* Patient under the influence of alcohol or psychotropic drugs
* Patient presenting a psychosis and/or a state of agitation, and/or a state of confusion.
* Patient presenting a hemodynamic, respiratory or neurological failure
* Patient with at least one of the following symptoms at the time of inclusion in the study: headache, dizziness, nausea, vomiting
* Persons benefiting from reinforced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection (guardianship and trusteeship) and finally patients in a vital emergency situation.
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy)
* Concurrent participation in another clinical research study whose objective is the evaluation of anxiety and/or pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Difference in anxiety level | 30 minutes
  Difference in anxiety level measured with a visual analog scale between T1 (before the analgesia-sedation procedure) and T4 (30 minutes after the procedure was performed, by asking the patient to rate the anxiety he or she felt during the procedure) during a technical procedure in traumatology in the emergency department in the VR group compared with the control group.
  The level of anxiety is measured with a visual analog scale (0: no anxiety, 10: maximum anxiety).

SECONDARY OUTCOMES:
Difference in pain intensity | 30 minutes
  The level of pain is measured with a visual analog scale (0: no pain, 10: maximum pain).
Doses of analgesics | During the procedure
  Total doses of analgesics used during a technical procedure performed in the context of trauma in the experimental group compared with the control group.
Occurrence of headache, nausea/vomiting, dizziness or confusional episode | During the procedure
  Tolerance assessed by looking for the occurrence of headache, nausea/vomiting, dizziness or confusional episode in both groups.
Evaluation of satisfaction | 30 minutes
  Comparison of the patient's level of satisfaction with pain and anxiety management between the two groups, assessed using a numerical scale ranging from 0 (not satisfied) to 10 (totally satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Poitiers, Poitiers, France